CLINICAL TRIAL: NCT04645849
Title: Feasibility Study on the Characterization of the Immune Profile of Young Patients After Treatment for Breast Cancer
Acronym: C-PiACs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.362; 2019-A02900-57 (Other: ID RCB)
Record Dates: First submitted 2020-06-15; First posted 2020-11-27 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: Immunity recovery; post treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples that will be destroyed after publications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A or "End of treatment": 16 patients recruited at the end of breast cancer treatment and followed during 9 months
  Interventions: Biological: Immunomonitoring
- Cohort B or "Diagnosis": Patients recruited at breast cancer before any treatment: one blood sample to provide comparative values.
  Interventions: Biological: Immunomonitoring

INTERVENTIONS:
Biological: Immunomonitoring — 16 patients will be recruited at the end of treatment: an immunoprofiling analysis will be performed out of a blood sample about 1 month, 5 months and 9 months after treatment.
  8 patients will be recruited at diagnosis: a immune profile analysis will be performed before the start of treatment. This will give comparative values for the immune system cells and molecules.

SUMMARY:
This study aim to determine kinetic of post treatment recovery/variation of a panel of innate and adaptative immune system cells and molecules.

The results should allow to determine the optimal post treatment immunomonitoring timing and panel to be used for future studies.

DETAILED DESCRIPTION:
There is a complexe interaction between tumor cells ans host immunity. Immunity system (IS) is clearly involved in cancer developement control, and it is suggested that it could participate to the response to anti cancer treatment.

There is however no validated immunomonitoring strategy to allow a reliable patient's immune status along time, and particularly after treatment.There are scarce existing information on immunologic reconstitution profile recovery after treatment.

This study aim to perform immunomonitoring in young patients with cancer to describe kinetic of recovery/variation of a panel of innate and adaptative immune system cells and molecules, selected by their potential relevance according to literature.

The concerned population are young women (˂40 yo) with breast cancer.

There will be 2 patients cohorts A or "End of treatment" : patients recruited at the end of treatment (study cohort) B or "Diagnosis" : Patients recruited at diagnosis (reference values)

This study should contribute to give sufficient data to determine the pertinent timing and cells/molecules panel to evaluate immunity profiling after treatment.

These results could be used for further studies.

ELIGIBILITY:
Inclusion Criteria:

* Women with Breast cancer at initial diagnosis OR at the end of treatment
* Chemotherapy planned or performed in the treatment plan
* Patient not opposed to participate to the present study
* Affiliated to a French social security scheme.

Exclusion Criteria:

* metastatic breast cancer
* pregnant or breastfeeding woman
* Treatment with monoclonal antibodies or immunotherapy
* Immunosuppressive therapy
* Thymus irradiation
* Chronic infection in progress
* Inborn or acquired disease (other than breast cancer) impacting the immune system (SAA, Lupus…)
* Subject under guardianship or deprived of liberty

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women with breast cancer and systemic treatments planed or done aged 18 to 39
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Identification of the relevant biological parameters of the innate / adaptive immune system | 15 months
  Analysis of immune profile implies to evaluate changes of about 30 distinct immune cell (sub)types with their activation markers. These analyses are conducted at 3 time points for cohort "A or End of treatment" (1, 5, 9 months) and once for cohort "B or Diagnosis" before treatment start :
  -% and counts of immune cell populations (B-lymphocytes, T-lymphocytes, dendritic cells)
  * activation levels of cell subpopulations
  * Secretion of cytokines after activation
  * Determination of cytokines and chemokines after activation (picograms/ml) Description of the evolution of the parameters measured for cohort "A or End of treatment" with comparison to normal values (data from the EFS cohort and from cohort "B or Diagnosis") Analysis of the reconstitution kinetic should allow us to determine wich biological parameters (immune cell (sub)types and their activation markers) will be most relevant to study immune profile reconstitution for further studies.

SECONDARY OUTCOMES:
Analysis feasibility | 15 months
  number of samples analysed versus planned, quality of the results
Immunity Cells and molecules kinetic analysis | 15 months
  The objective is to determine the best moment for analysis of immune system reconstitution (cf outcome 1 measures) For each patient, and each immune system marker tested (cells/molecules): kinetic analysis of return to values comparable to reference values (data from the EFS = french blood establishment and the 8 patients tested before the start of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Leila Gofti-Laroche, PharmD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No